CLINICAL TRIAL: NCT07162441
Title: A Two-arm, Open-label, Single-sequence, Multiple-dose, Cross-over Study to Evaluate the Pharmacokinetic Interaction and the Safety of UIC202502 and UIC202505 in Healthy Adult Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-UI113-101
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: treatment A; Drug: treatment C
- Arm B (Experimental)
  Interventions: Drug: treatment B; Drug: treatment C

INTERVENTIONS:
Drug: treatment A — UIC202502 1 Tab/day for 7 days
  Arms: Arm A
Drug: treatment B — UIC202505 1 Tab/day for 7 days
  Arms: Arm B
Drug: treatment C — UIC202502+UIC202505 2 Tab/day for 7 days

SUMMARY:
This study is open-label, multiple-dose, two-intervention group, single-sequence, crossover design to compare the safety and pharmacokinetics of UIC202502 and UIC202505 when administered alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 19 years or older at the time of screening.
* Subjects with a body weight greater than 50 kg (≥45 kg for females) and a body mass index (BMI) between 18.0 and 30.0 kg/m² at screening.

(BMI (kg/m²) = weight (kg) / height (m)²)

* Subjects with no clinically significant congenital or chronic diseases, pathological symptoms or findings at screening.
* Subjects determined by the principal investigator to be suitable for diagnostic procedures and electrocardiogram assessments
* Subjects who agree to use an effective method of contraception (excluding hormonal agents) recognized as appropriate in clinical trials from the first administration of the investigational drug until 14 days after the last administration, together with their spouse or partner.
* Subjects who have provided written informed consent after receiving a full explanation and demonstrating an understanding of the purpose, procedures, and characteristics of this clinical trial and the investigational drug.

Exclusion Criteria:

* Subjects with clinically significant diseases or a history of conditions involving the digestive, cardiovascular, endocrine, respiratory, hematologic/oncologic infectious, renal/genitourinary, psychiatric/neurologic, musculoskeletal, immune, otorhinolaryngologic, dermatologic, or ophthalmologic systems.
* Subjects with a history of gastrointestinal surgery (excluding simple appendectomy or hernia repair) or gastrointestinal disease that may affect drug absorption.
* Subjects who have taken drugs that induce or inhibit drug-metabolizing enzymes (e.g., barbiturates) within 1 month before the first dose, or drugs that may interfere with this clinical trial within 10 days before the first dose
* Subjects who have participated in another clinical trial or bioequivalence study and received an investigational drug within 6 months before the first administration.
* Subjects who have donated whole blood or blood components within 2 weeks, or received a blood transfusion within 4 weeks before the first administration.
* Subjects who meet any of the following criteria within 1 month before the first dose:

  * Average alcohol consumption exceeding 21 drinks/week for men
  * Average alcohol consumption exceeding 14 drinks/week for women

    (1 drink = 50 mL soju, 30 mL liquor, or 250 mL beer)
  * Smoking more than 20 cigarettes/day on average
* Subjects judged by the principal investigator to be unsuitable for participation in this clinical trial for any reason other than the above selection or exclusion criteria.
* Female subjects who are pregnant, suspected of being pregnant, or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
AUCτ | 0 to 24hr
  Evaluation PK
Cmax,ss | 0 to 24hr
  Evaluation PK

CONTACTS AND LOCATIONS:
Locations (1):
- H plus Yangji Hospital, Seoul, Gwanak-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided